CLINICAL TRIAL: NCT00460031
Title: Phase II Trial to Assess the Activity of Ketoconazole Plus Lenalidomide in Patients With Prostate Cancer Progressive After Androgen Deprivation
Brief Title: Treating Patients With Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE12805
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ketoconazole; 1-methyl-4-(1-naphthylvinyl)piperidine; Lenalidomide; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketoconazole Plus Lenalidomide (Experimental)
  Interventions: Drug: ketoconazole; Drug: lenalidomide; Drug: therapeutic hydrocortisone

INTERVENTIONS:
Drug: ketoconazole — 400 tid
  Other Names: held for toxicity, missed days of therapy are not made up.
Drug: lenalidomide — Lenalidomide will be administered daily at a dose of 25mg po qd on days 1-21 of the cycle.
Drug: therapeutic hydrocortisone — 20mg qam 10mg qhs

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Drugs, such as ketoconazole, may stop the adrenal glands from making androgens. Lenalidomide may stop the growth of prostate cancer by blocking blood flow to the tumor. Giving ketoconazole and hydrocortisone together with lenalidomide may be an effective treatment for prostate cancer.

PURPOSE: This phase II trial is studying how well giving ketoconazole and hydrocortisone together with lenalidomide works in treating patients with prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response frequency in patients with hormone-refractory progressive prostate cancer treated with ketoconazole, hydrocortisone, and lenalidomide.

Secondary

* Determine the effect of this regimen on time to clinical progression in these patients.
* Determine the safety of this regimen in these patients.
* Determine the effects of this regimen on serum cytokines, including tumor necrosis factor-alpha, basic fibroblast growth factor, plasma soluble interleukin (IL)-2 receptor, IL-8, and IL-12, as well as serum vascular endothelial growth factor levels in these patients.
* Determine the co-stimulatory effects of this regimen on dendritic cells and CD4-positive, CD25-positive, T-regulatory cells in these patients.

OUTLINE: This is a nonrandomized, open-label study.

Patients receive oral ketoconazole 3 times daily and oral hydrocortisone twice daily on days 1-28 and oral lenalidomide once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically during study for evaluation of prostate cancer-specific immune response. Blood samples are assessed by serum analysis, flow cytometry, real-time PCR, and enzyme-linked immunosorbent assay techniques to detect and quantify different cytokines, antiangiogenic markers, dendritic cells, and specific T-regulatory cells.

After completion of study therapy, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
PATIENTS WITH PROSTATE CANCER PROGRESSIVE AFTER ANDROGEN DEPRIVATION Inclusion Criteria Understand and voluntarily sign an informed consent form. Age 18 years at the time of signing the informed consent form. Histologically confirmed adenocarcinoma of the prostate. Testosterone less than 50 ng/dL. Patients must continue primary androgen deprivation with an LHRH analogue if they have not undergone orchiectomy. All previous cancer therapy, including radiation, and surgery, must have been discontinued at least 4 weeks prior to receive first dose of study drug.

Progressive disease after androgen deprivation.

Exclusion Criteria Prior systemic chemotherapy for hormone refractory prostate cancer. Prior neoadjuvant and adjuvant chemotherapy are allowed when completed at least 12 months prior to enrollment.

Prior ketoconazole, aminoglutethimide or corticosteroids for the treatment of progressive prostate cancer.

Prior immunotherapy including, but not limited to, vaccines, Thalidomide, and or Lenalidomide like agents.

Supplements or complementary medicines/botanicals are not permitted while on protocol therapy, except for any combination of the following:

conventional multivitamin supplements selenium lycopene soy supplements Patients should review the label with their doctor prior to enrollment, and discontinue disallowed agents prior to study enrollment Serious intercurrent infections or non-malignant medical illnesses including autoimmune disorders that are uncontrolled.

Psychiatric illnesses/social situations that would limit compliance with protocol requirements.

Evidence of CNS (brain or Leptomeningeal) metastases or large pleural/pericardial effusions.

Known contraindication to receive Ketoconazole or Lenalidomide Concurrent use of ketoconazole with statin compounds is absolutely contraindicated. Thus, patients receiving Statin drugs (fluvastatin, atorvastatin, and simvastatin) should discontinue them for at least 7 days before starting ketoconazole.

Patients taking astemizole, terfenadine, or cisapride, rifampin or isoniazid are not eligible, unless they agreed to completely discontinue those agents. In that case, any of these agents should be discontinued at least 7 days prior to start therapy with Ketoconazole.

Use of any other experimental drug or therapy within 28 days of baseline. Known hypersensitivity to thalidomide or its analogues. Any prior use of Lenalidomide. Known positive for HIV or infectious hepatitis, type A, B or C. Disease free of prior malignancies for 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the breast.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Matthew M. Cooney, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (6):
- United States (6):
  - Lake/University Seidman Cancer Center, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Barata PC, Cooney M, Mendiratta P, Tyler A, Dreicer R, Garcia JA. Ketoconazole plus Lenalidomide in patients with Castration-Resistant Prostate Cancer (CRPC): results of an open-label phase II study. Invest New Drugs. 2018 Dec;36(6):1085-1092. doi: 10.1007/s10637-018-0660-3. Epub 2018 Sep 6. PMID 30191523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty seven (37) patients were screened from Cleveland Clinic and University Hospitals in the Cleveland area from February 2007 to April 2009.Three patients were not eligible.
Groups:
- Ketoconazole Plus Lenalidomide: Ketoconazole will be administered daily on days 1-28 of the cycle at a dose of 400mg po tid with hydrocortisone 20mg po every morning and 10mg po at bedtime. Hydrocortisone will be given on a continuous basis. Lenalidomide will be administered daily at a dose of 25mg po qd on days 1-21 of the cycle.
Period: Overall Study
Arm/Group | Ketoconazole Plus Lenalidomide
Started | 34
Completed | 23
Not Completed | 11
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 5
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketoconazole Plus Lenalidomide
Number analyzed (Participants) | 34
Age, Customized [Number; unit: participants]
  40-49 years | 2
  50-59 years | 5
  60-69 years | 10
  70-79 years | 11
  80-89 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Partial Response, Progressive Disease, or Stable Disease Based on Prostate-Specific Antigen (PSA) or Measurable Disease
Description: Patients will be evaluated for clinical benefit monthly with PSA values.Patients who are benefiting from treatment are eligible for additional cycles of treatment. Thereafter, therapy will continue until criteria for progressive disease are met. Response is based on the RECIST criteria from the National Cancer institute. Complete Response (CR) disappearance of all target lesions; Partial Response (PR) >= 30% decrease in the sum of the longest diameter of target lesions from baseline; Progressive Disease (PD) >= increase in the sum of the longest diameter of target lesions from baseline; Stable Disease (SD) neither sufficient for partial response nor sufficient increase for progressive disease.
Time Frame: 28 days
Population: All patients who completed the study
Measure: Number; unit: participants
Arm/Group | Ketoconazole Plus Lenalidomide
Number analyzed (Participants) | 23
participants
  Partial Response | 7
  Progressive Disease | 7
  Stable Disease | 9

2. Secondary Outcome: Time to Progression
Description: as for outcome 1
Time Frame: One year (12 months) after start of treatment
Population: Patients with disease progression
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ketoconazole Plus Lenalidomide
Number analyzed (Participants) | 7
Months | 3 [-1.52 to 7.52]

3. Secondary Outcome: Number of Patients With Grade 3 and 4 Toxicity as Assessed by NCI CTCAE v3.0
Description: Patients will be evaluated for toxicity every 2 weeks during the first cycle. Thereafter, evaluations will be done every 28 days or more frequently if clinically indicated.
Time Frame: Up to 30 days after discontinuation of treatment
Population: All patients who received at least one treatment in the study
Measure: Number; unit: participants
Arm/Group | Ketoconazole Plus Lenalidomide
Number analyzed (Participants) | 34
participants | 19

4. Secondary Outcome: Change in Immune Response From Baseline
Description: The pattern of immune response by assessing T cell and dendritic cell markers, specifically by measuring the levels of CD4+ FoxP3+ Regulatory T cells
Time Frame: Week 8
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: cells/ul
Arm/Group | Ketoconazole Plus Lenalidomide
Number analyzed (Participants) | 23
cells/ul | 0.18 (0.31)

5. Secondary Outcome: Ratio of Change in Immune Response From Baseline
Description: The pattern of immune response by assessing T cell and dendritic cell markers, specifically by measuring the ratio of BDCA-2 to BDCA-1 cells
Time Frame: Week 8
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ketoconazole Plus Lenalidomide
Number analyzed (Participants) | 23
ratio | -0.39 (1.44)

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Ketoconazole Plus Lenalidomide
Serious Adverse Events (participants affected / at risk) | 12/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketoconazole Plus Lenalidomide (N=34)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Cardiovascular/Arrhythmia (Cardiac disorders) | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 1
Cardiovascular/General (Cardiac disorders) | 2
Edema (General disorders) | 1
Coagulation (Blood and lymphatic system disorders) | 1
Constitutional Symptoms (General disorders) | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
dehydration (Gastrointestinal disorders) | 1
Diarrhea patients without colostomy (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Bilirubin (Investigations) | 1
Liver dysfunction (Hepatobiliary disorders) | 1
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 1
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 1
Infection/Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1
Dizziness/lightheadedness (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Fatigue (Lethargy, malaise, asthenia) (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketoconazole Plus Lenalidomide (N=34)
"Fatigue (lethargy, malaise, asthenia)" (General disorders) | 27 (50)
General Disorders (General disorders) | 5 (7)
"Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L)" (General disorders) | 3 (3)
Weight loss (General disorders) | 3 (10)
"Rigors, chills" (General disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 14 (18)
Anorexia (Gastrointestinal disorders) | 10 (12)
Constipation (Gastrointestinal disorders) | 10 (12)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 7 (9)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 5 (7)
Dyspepsia/heartburn (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 2 (2)
Mouth dryness (Gastrointestinal disorders) | 2 (2)
Hemoglobin (Investigations) | 18 (38)
Lymphopenia (Investigations) | 17 (61)
Platelets (Blood and lymphatic system disorders) | 13 (37)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 12 (47)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 10 (30)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16 (28)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (14)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 14 (34)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (14)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 8 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (7)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Bicarbonate (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Edema (General disorders) | 13 (18)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 3 (3)
Thrombosis/embolism (Vascular disorders) | 3 (4)
Cardiovascular/General (Vascular disorders) | 2 (2)
Alkaline phosphatase (Investigations) | 13 (19)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 13 (19)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 11 (17)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (21)
Bilirubin (Investigations) | 2 (4)
Dizziness/lightheadedness (Nervous system disorders) | 9 (12)
Insomnia (Psychiatric disorders) | 5 (5)
Neuropathy-sensory (Nervous system disorders) | 4 (5)
Mood alteration-depression (Nervous system disorders) | 3 (3)
Neurology-Other (Nervous system disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 12 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine (Investigations) | 10 (20)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Urinary discoloration (Renal and urinary disorders) | 2 (2)
Pain (General disorders) | 11 (23)
Chest pain (non-cardiac and non-pleuritic) (Cardiac disorders) | 3 (3)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (15)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 6 (6)
Infection/Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (10)
Infection without neutropenia (Infections and infestations) | 5 (6)
Dry eye (Eye disorders) | 4 (6)
Vision-blurred vision (Eye disorders) | 4 (6)
Ocular/Visual (Eye disorders) | 2 (2)
Vision-flashing lights/floaters (Eye disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hemorrhage (Vascular disorders) | 4 (5)
"Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip)" (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Allergy (Immune system disorders) | 2 (2)
Hot flashes/flushes (Endocrine disorders) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Coagulation (Blood and lymphatic system disorders) | 3 (4)
Auditory/Hearing (Ear and labyrinth disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes